CLINICAL TRIAL: NCT03752021
Title: The Endocannabinoid System in Human Gestational Tissues in Labor
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00051905
Record Dates: First submitted 2018-11-21; First posted 2018-11-23 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-06

CONDITIONS: Labor
Keywords: Endocannabinoid System; Human Gestational Tissues; Labor; Cesarean Section

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — A sample of the uterus will be removed at the existing incision made by your doctors. The uterine segment (sample) will be 2 inches in length and 0.5 inches in width. The placenta and the attached membranes will also be collected for the study. The uterine incision will be repaired in the standard fashion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Laboring Subjects: Subjects with a planned cesarean delivery who labor prior to their scheduled date or those who are in labor and require an unplanned but non-emergent cesarean delivery. These subjects will be approached upon admission to the study facility by the researcher for potential enrollment to allow adequate time to consider participation, ask questions, provide consent, and prior to procedure (Myometrial Sampling).
  Interventions: Procedure: Myometrial Sampling
- Non Laboring Subjects: Subjects with a planned cesarean delivery will be approached by the researcher during prenatal visits or at the study facilities prior to planned procedure (Myometrial Sampling)
  Interventions: Procedure: Myometrial Sampling

INTERVENTIONS:
Procedure: Myometrial Sampling — A myometrial sample will be obtained at the time of cesarean delivery. Sample will be obtained from the superior edge of the existing lower uterine segment incision and will be 2 inches in length and 0.5 inches in width. The uterine incision will be repaired in a standard two-layer closure. If a classical cesarean (vertical) uterine incision is deemed necessary and is performed by the surgical team, a sample of the same size will be taken parallel to the incision at the existing edge. The classical uterine incision will be closed utilizing the standard layered technique.
  Placenta and gestational membrane tissue will be obtained after placental delivery. The entire placenta and attached gestational membranes will be collected if not being sent for pathologic review

SUMMARY:
The purpose of this research study is to determine if the endocannabinoid (a biological system) plays a role in the labor process.

DETAILED DESCRIPTION:
This is a pilot study to determine the feasibility of identification and quantification of various components of the endocannabinoid system in the labored versus non-labored myometrium, placenta and gestational membranes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women ages > 18 years old
* Pregnant women 22 weeks, 0 days through 42 weeks, 0 days gestation undergoing cesarean section
* Singleton gestation

Exclusion Criteria:

* Cannabinoid use during pregnancy
* Illicit drug use during pregnancy
* Nonsteroidal anti-inflammatory drug use within 7 days of cesarean section
* Maternal comorbidities including pre-existing diabetes, pre-existing hypertension, hypertensive disorders of pregnancy (preeclampsia, eclampsia), epilepsy currently being treated with antiepileptic medication, intraamniotic infection
* Uterine abnormalities
* Fetal anomalies
* Drug use or dependency

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: * A total of 20 subjects will be enrolled in the pilot study
  * 10 laboring subjects
  * 10 non-laboring subjects
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Presence of CB1 receptor protein | At the time of C-section
  Identification of CB1 receptor protein interacting protein (CRIP) in gestational membranes, placenta, and myometrium
Presence of CB2 receptor protein | At the time of C-section
  Identification of CB2 receptor protein interacting protein (CRIP) in gestational membranes, placenta, and myometrium
Presence of cannabinoid receptor | At the time of C-section
  Identification of cannabinoid receptor interacting protein (CRIP) in gestational membranes, placenta, and myometrium
Levels of CB1 receptor protein | At the time of C-section
  Quantification of levels of CB1 receptor protein interacting protein (CRIP) in gestational membranes, placenta, and myometrium. A statistical comparison between groups will be performed.
Levels of CB2 receptor protein | At the time of C-section
  Quantification of CB2 receptor protein interacting protein (CRIP) in gestational membranes, placenta, and myometrium. A statistical comparison between groups will be performed.
Levels of cannabinoid receptor | At the time of C-section
  Quantification of cannabinoid receptor interacting protein (CRIP) in gestational membranes, placenta, and myometrium. A statistical comparison between groups will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa L Kozakiewicz, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina

REFERENCES:
- [Background] Navathe R, Berghella V. Tocolysis for Acute Preterm Labor: Where Have We Been, Where Are We Now, and Where are We Going? Am J Perinatol. 2016 Feb;33(3):229-35. doi: 10.1055/s-0035-1571147. Epub 2016 Jan 25. PMID 26808195
- [Background] Goldenberg RL, Culhane JF, Iams JD, Romero R. Epidemiology and causes of preterm birth. Lancet. 2008 Jan 5;371(9606):75-84. doi: 10.1016/S0140-6736(08)60074-4. PMID 18177778
- [Background] Matsuda LA, Lolait SJ, Brownstein MJ, Young AC, Bonner TI. Structure of a cannabinoid receptor and functional expression of the cloned cDNA. Nature. 1990 Aug 9;346(6284):561-4. doi: 10.1038/346561a0. PMID 2165569
- [Background] Howlett AC, Bidaut-Russell M, Devane WA, Melvin LS, Johnson MR, Herkenham M. The cannabinoid receptor: biochemical, anatomical and behavioral characterization. Trends Neurosci. 1990 Oct;13(10):420-3. doi: 10.1016/0166-2236(90)90124-s. PMID 1700516
- [Background] Paria BC, Song H, Wang X, Schmid PC, Krebsbach RJ, Schmid HH, Bonner TI, Zimmer A, Dey SK. Dysregulated cannabinoid signaling disrupts uterine receptivity for embryo implantation. J Biol Chem. 2001 Jun 8;276(23):20523-8. doi: 10.1074/jbc.M100679200. Epub 2001 Mar 8. PMID 11279117
- [Background] Paria BC, Dey SK. Ligand-receptor signaling with endocannabinoids in preimplantation embryo development and implantation. Chem Phys Lipids. 2000 Nov;108(1-2):211-20. doi: 10.1016/s0009-3084(00)00197-3. PMID 11106792
- [Background] Das SK, Paria BC, Chakraborty I, Dey SK. Cannabinoid ligand-receptor signaling in the mouse uterus. Proc Natl Acad Sci U S A. 1995 May 9;92(10):4332-6. doi: 10.1073/pnas.92.10.4332. PMID 7753807
- [Background] Schmid PC, Paria BC, Krebsbach RJ, Schmid HH, Dey SK. Changes in anandamide levels in mouse uterus are associated with uterine receptivity for embryo implantation. Proc Natl Acad Sci U S A. 1997 Apr 15;94(8):4188-92. doi: 10.1073/pnas.94.8.4188. PMID 9108127
- [Background] Paria BC, Wang H, Dey SK. Endocannabinoid signaling in synchronizing embryo development and uterine receptivity for implantation. Chem Phys Lipids. 2002 Dec 31;121(1-2):201-10. doi: 10.1016/s0009-3084(02)00156-1. PMID 12505701
- [Background] Dennedy MC, Friel AM, Houlihan DD, Broderick VM, Smith T, Morrison JJ. Cannabinoids and the human uterus during pregnancy. Am J Obstet Gynecol. 2004 Jan;190(1):2-9; discussion 3A. doi: 10.1016/j.ajog.2003.07.013. PMID 14749627
- [Background] Park B, Gibbons HM, Mitchell MD, Glassa M. Identification of the CB1 cannabinoid receptor and fatty acid amide hydrolase (FAAH) in the human placenta. Placenta. 2003 May;24(5):473-8. doi: 10.1053/plac.2002.0926. PMID 12744923
- [Background] Wang H, Xie H, Dey SK. Loss of cannabinoid receptor CB1 induces preterm birth. PLoS One. 2008 Oct 3;3(10):e3320. doi: 10.1371/journal.pone.0003320. PMID 18833324
- [Background] Habayeb OM, Taylor AH, Evans MD, Cooke MS, Taylor DJ, Bell SC, Konje JC. Plasma levels of the endocannabinoid anandamide in women--a potential role in pregnancy maintenance and labor? J Clin Endocrinol Metab. 2004 Nov;89(11):5482-7. doi: 10.1210/jc.2004-0681. PMID 15531501
- [Background] Costa MA, Fonseca BM, Keating E, Teixeira NA, Correia-da-Silva G. 2-arachidonoylglycerol effects in cytotrophoblasts: metabolic enzymes expression and apoptosis in BeWo cells. Reproduction. 2014 Feb 3;147(3):301-11. doi: 10.1530/REP-13-0563. Print 2014 Mar. PMID 24324206
- [Background] Chiossi G, Costantine MM, Bytautiene E, Kechichian T, Hankins GD, Sbrana E, Saade GR, Longo M. The effects of prostaglandin E1 and prostaglandin E2 on in vitro myometrial contractility and uterine structure. Am J Perinatol. 2012 Sep;29(8):615-22. doi: 10.1055/s-0032-1311986. Epub 2012 May 25. PMID 22639355
- [Background] Chioss G, Costantine MM, Bytautiene E, Betancourt A, Hankins GD, Saade GR, Longo M. In vitro myometrial contractility profiles of different pharmacological agents used for induction of labor. Am J Perinatol. 2012 Oct;29(9):699-704. doi: 10.1055/s-0032-1314891. Epub 2012 May 29. PMID 22644831
- [Background] Luckas MJ, Wray S. A comparison of the contractile properties of human myometrium obtained from the upper and lower uterine segments. BJOG. 2000 Oct;107(10):1309-11. doi: 10.1111/j.1471-0528.2000.tb11626.x. PMID 11028587
- [Background] Moynihan AT, Smith TJ, Morrison JJ. The relaxant effect of nifedipine in human uterine smooth muscle and the BK(Ca) channel. Am J Obstet Gynecol. 2008 Feb;198(2):237.e1-8. doi: 10.1016/j.ajog.2007.08.074. PMID 18226634
- [Background] Quenby S, Matthew A, Zhang J, Dawood F, Wray S. In vitro myometrial contractility reflects indication for caesarean section. BJOG. 2011 Nov;118(12):1499-506. doi: 10.1111/j.1471-0528.2011.03064.x. Epub 2011 Jul 27. PMID 21790954
- [Derived] Kozakiewicz ML, Zhang J, Leone-Kabler S, Yamaleyeva LM, McDonald AG, Brost BC, Howlett AC. Differential Expression of CB1 Cannabinoid Receptor and Cannabinoid Receptor Interacting Protein 1a in Labor. Cannabis Cannabinoid Res. 2022 Jun;7(3):279-288. doi: 10.1089/can.2020.0107. Epub 2021 Apr 16. PMID 33998898